CLINICAL TRIAL: NCT02242695
Title: Comparative Study of the Efficacy of 10.0 mg Dequalinium Chloride (Fluomizin®) and 100 mg Clotrimazole (Canesten®) for the Treatment of Vulvovaginal Candidiasis
Brief Title: Comparative Efficacy Study of 10 mg Dequalinium Chloride (Fluomizin) in the Treatment of Vulvovaginal Candidiasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medinova AG (Industry)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Flu-380112
Record Dates: First submitted 2013-10-23; First posted 2014-09-17 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2015-07

CONDITIONS: Vulvovaginal Candidiasis
Keywords: vulvovaginal candidiasis; vulvovaginal candidosis; mycotic vaginal infection; dequalinium chloride; Fluomizin; clotrimazole; canesten
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluomizin vaginal tablets (Experimental): Fluomizin vaginal tablets containing 10mg dequalinium chloride once daily for 6 days and one placebo vaginal tablet on day 7
  Interventions: Drug: Fluomizin vaginal tablets
- Canesten vaginal tablets (Active Comparator): Canesten vaginal tablets containing 100mg clotrimazole once daily for 7 days
  Interventions: Drug: Canesten vaginal tablets

INTERVENTIONS:
Drug: Fluomizin vaginal tablets — One vaginal tablet for 6 days and 1 placebo tablet on day 7
  Other Names: 10 mg dequalinium chloride vaginal tablets; Donaxyl vaginal tablets; Naxyl vaginal tablets
  Arms: Fluomizin vaginal tablets
Drug: Canesten vaginal tablets — one vaginal tablet for 7 days
  Other Names: 100mg clotrimazole vaginal tablets
  Arms: Canesten vaginal tablets

SUMMARY:
A clinical study to compare the clinical efficacy of vaginal tablets containing 10mg dequalinium chloride (Fluomizin) with the clinical efficacy of 100mg clotrimazole in patients suffering from vulvovaginal candidiasis, to assess safety of the two medications during the treatment, and to evaluate women's satisfaction with the two treatments.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and symptoms of vulvovaginal candididiasis as Total Severity Score, Total Severity Score of at least 4 (0-15: vaginal itching (0-3), vaginal burning or soreness (0-3), abnormal vaginal discharge (0-3),vulvo/vaginal erythema or edema(0-3), vulvar excoriation or fissure formation (0-3).
* Direct microscopy (Wet smear) positive for yeast forms (hyphae/pseudohyphae) or budding yeasts.
* normal vaginal pH (higher than 4.5) at baseline.
* Women aged 18 - 45 years old.
* Women can comply with all clinical trial instructions, and can return to all follow-up visits.
* Signed Written Informed Consent to participate in this study.

Exclusion Criteria:

* Recurrent vulvovaginal candidiasis(4 episodes of VVC in the last 12 months).
* Women with other cause of vaginal infections, e.g. bacterial vaginosis, aerobic vaginitis, trichomoniasis, and mixed infections
* Women using oral or vaginal antifungals within 2 weeks prior to enrolment and during the study.
* Women using any intra-vaginal products, also vaginal douches containing soaps and other anionic, surface-active substances, within 2 weeks prior to enrolment and during the study.
* Women using any antibiotic or anti-infective within 2 weeks prior to enrolment.
* Cervicitis, abnormal PAP smear in the last 6 month.
* Severe systemic diseases (HIV infection, diabetes mellitus, cancer, tuberculosis, autoimmune diseases, severe psychiatric conditions, etc.).
* Women with confirmed Neisseria gonorrhoea or Chlamydia trachomatis.
* Women having menstruation bleeding at enrolment.
* Known or suspected hypersensitivity to one of the study medications, inclusive their excipients.
* Participation of patient in another investigational drug study concomitantly or within 30 days prior to entry in the study.
* Patient is relative of, or staff directly reporting to, the investigator.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate | Control 1 at day 4 after therapy end
  Clinical cure rate is defined as Total Severity Score (TSC) ≤ 2

SECONDARY OUTCOMES:
Microbiological cure rate | Control 1 at 4 days after therapy end
  Negative microscopy for showing yeast forms (hyphae/pseudohyphae) or budding yeasts and Negative Candida culture
Therapeutic cure rate | Control 1 at 4 days after therapy end
  Clinically and microbiologically cured
Individual clinical signs and symptoms | Control 1 at 4 days after therapy end
  4-point rating scale for vaginal itching, vaginal burning or soreness, vulvo/vaginal erythema or edema, and vulvar excoriation ofr fissure formation
Presence of dyspareunia | Control 1 at 4 days after therapy end
  yes/no
Direct microscopy (wet smear) | Control 1 at 4 days after therapy end
  Presence or absence of Candida hyphea or spores
vaginal pH | Control 1 at 4 days after therapy end
Candida culture | Control 1 at 4 days after therapy end
  positive / negative for Candida spp
Global assessment of efficacy | Control 1 at 4 days after therapy end
  4-point rating scale assessed by investigator and patient
Patient Satisfaction | Control 1 at 4 days after therapy end
  presence of vaginal discomfort, increased discharge, burning sensation
Adverse event | Control 1 at 4 days after therapy end
  Number of participants experiencing an adverse event
Global assessment of tolerability | Control 1 at 4 days after therapy end
  4-point rating scale by investigator and patient
Clinical cure rate | Control 2 at 6 weeks after therapy end
  Clinical cure rate defined as Total Symptom Score TSC ≤ 2
Presence of external dysuria | Control 1 at 4 days after therapy end
  yes/no
Microbiological cure rate | Control 2 at 6 weeks after therapy end
  Negative microscopy for showing yeast forms (hyphae/pseudohyphae) or budding yeasts and Negative Candida culture
Therapeutic cure rate | Control 2 at 6 weeks after therapy end
  Clinically and microbiologically cured
Individual clinical signs and symptoms | Control 2 at 6 weeks after therapy end
  4-point rating scale for vaginal itching, vaginal burning or soreness, vulvo/vaginal erythema or edema, and vulvar excoriation ofr fissure formation
Presence of dyspareunia | Control 2 at 6 weeks after therapy end
  yes/no
Direct microscopy (wet smear) | Control 2 at 6 weeks after therapy end
  Presence or absence of Candida hyphea or spores
vaginal pH | Control 2 at 6 weeks after therapy end
Candida culture | Control 2 at 6 weeks after therapy end
  positive / negative for Candida spp
Global assessment of efficacy | Control 2 at 6 weeks after therapy end
  4-point rating scale assessed by investigator and patient
Patient Satisfaction | Control 2 at 6 weeks after therapy end
  presence of vaginal discomfort, increased discharge, burning sensation
Adverse event | Control 2 at 6 weeks after therapy end
  Number of participants experiencing an adverse event
Global assessment of tolerability | Control 2 at 6 weeks after therapy end
  4-point rating scale by investigator and patient
Presence of external dysuria | Control 2 at 6 weeks after therapy end
  yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Manopchai Thamkhantho, Prof MD, Principal Investigator — Siriraj Gynaecologic ID and Female STD Unit, Mahidol University
Locations (1):
- Siriraj Gynaecologic ID and Female STD Unit, Department of Obstetrics & Gynaecology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok Noi District, Thailand

REFERENCES:
- [Derived] Thamkhantho M, Chayachinda C. Vaginal tablets of dequalinium chloride 10 mg versus clotrimazole 100 mg for vaginal candidiasis: a double-blind, randomized study. Arch Gynecol Obstet. 2021 Jan;303(1):151-160. doi: 10.1007/s00404-020-05784-z. Epub 2020 Sep 17. PMID 32940765